CLINICAL TRIAL: NCT02548910
Title: The PRICE Trial: Phlebotomy Resulting in Controlled Hypovolemia to Prevent Blood Loss in Major Hepatic Resections
Brief Title: Phlebotomy to Prevent Blood Loss in Major Hepatic Resections
Acronym: PRICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3588
Record Dates: First submitted 2015-07-23; First posted 2015-09-14 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Liver Neoplasms; Hepatectomy
MeSH Terms: conditions — Liver Neoplasms | interventions — Phlebotomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phlebotomy (Experimental): For patients randomized to phlebotomy, the intervention will consist of the standard of care (low CVP surgery), plus whole blood phlebotomy. Blood will be collected in citrated whole blood collection bag.
  Interventions: Procedure: Phlebotomy; Device: Citrated whole blood collection bag
- Control (No Intervention): Standard of care (low CVP surgery). In this arm, standard anesthesia will be maintained.

INTERVENTIONS:
Procedure: Phlebotomy — A central venous catheter will be inserted for every patient to measure central venous pressure, as is the standard of care in elective liver surgery. Strict aseptic technique will be maintained. A total volume of whole blood of 7-10 mL per kg of body weight will be removed, as tolerated. The volume of removed blood will not be replaced by intravenous fluid administration. Collected blood will be transfused back at the end of the liver parenchymal transection, or within 8 hours of collection.
  Arms: Phlebotomy
Device: Citrated whole blood collection bag — Transfusion Medicine will send the requested number of whole blood collection bags labelled with the patient's name and MRN. These whole blood collection bags are used in standard practice for collection of whole blood.
  Arms: Phlebotomy

SUMMARY:
Major liver resection is associated with substantial intraoperative blood loss. Blood loss in elective liver surgery is a significant factor of perioperative morbidity and mortality, as well as possibly long-term oncologic outcome. The purpose of this study is to use whole blood phlebotomy to decrease the central venous pressure, resulting in a state of relative hypovolemia. It is hypothesized that this intervention will lead to a decrease in blood loss at the time of liver resection.

DETAILED DESCRIPTION:
Major liver resection is associated with significant intraoperative blood loss. Blood loss in elective liver surgery is a key determinant of perioperative morbidity and mortality, as well as possibly long-term oncologic outcome. Whole blood phlebotomy is a simple intervention, whose aim is to decrease the central venous pressure yielding a state of relative hypovolemia and thus lead to decreased blood loss. Small studies, mostly from the liver transplant literature, would suggest that phlebotomy with controlled hypovolemia can result in decreased blood loss and blood transfusion. Since blood loss is an important issue in liver surgery, and the benefits of phlebotomy and controlled hypovolemia are unknown in liver resection patients, a rigorously conducted trial in a representative population of patients undergoing liver resection is warranted, and feasible. In this proposal, it is hypothesized that by the use of phlebotomy and controlled hypovolemia, it is possible to decrease blood loss and blood transfusions. To test this hypothesis the investigators plan to randomly allocate participants to phlebotomy plus standard of care or to standard of care. Participants will be those patients undergoing elective major liver resection at the Ottawa Hospital for any indication. The primary outcome will be intraoperative blood loss. Secondary outcomes will include transfusion requirements, perioperative morbidity and mortality, safety, physiologic parameters, and feasibility elements. A total of 62 patients will be randomized. The efficacy of phlebotomy in terms of blood loss prevention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Any patient being considered for a major elective liver resection will be considered for trial enrollment. Patients who are undergoing a concurrent additional abdominal or thoracic procedure (eg. colonic resection) will also be included.

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Refusal of blood products
* Active cardiac conditions: unstable coronary syndromes, decompensated heart failure (NYHA functional class IV; worsening or new-onset heart failure), significant arrhythmias, severe valvular disease
* History of significant cerebrovascular disease
* Renal dysfunction (patients with an estimated GFR <60 mL/min)
* Abnormal coagulation parameters (INR >1.5 not on warfarin and/or platelets count <100 X109/L )
* Evidence of hepatic metabolic disorder (bilirubin >35 umol/L)
* Presence of active infection
* Preoperative autologous blood donation
* Hemoglobin <100 g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Martel, MD, MSc, FRCSC, FACS, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hashimoto T, Kokudo N, Orii R, Seyama Y, Sano K, Imamura H, Sugawara Y, Hasegawa K, Makuuchi M. Intraoperative blood salvage during liver resection: a randomized controlled trial. Ann Surg. 2007 May;245(5):686-91. doi: 10.1097/01.sla.0000255562.60215.3b. PMID 17457160
- [Background] Alkozai EM, Lisman T, Porte RJ. Bleeding in liver surgery: prevention and treatment. Clin Liver Dis. 2009 Feb;13(1):145-154. doi: 10.1016/j.cld.2008.09.012. PMID 19150318
- [Background] Huntington JT, Royall NA, Schmidt CR. Minimizing blood loss during hepatectomy: a literature review. J Surg Oncol. 2014 Feb;109(2):81-8. doi: 10.1002/jso.23455. Epub 2013 Oct 4. PMID 24449171
- [Background] McNally SJ, Revie EJ, Massie LJ, McKeown DW, Parks RW, Garden OJ, Wigmore SJ. Factors in perioperative care that determine blood loss in liver surgery. HPB (Oxford). 2012 Apr;14(4):236-41. doi: 10.1111/j.1477-2574.2011.00433.x. Epub 2012 Feb 28. PMID 22404261
- [Background] Jarnagin WR, Gonen M, Fong Y, DeMatteo RP, Ben-Porat L, Little S, Corvera C, Weber S, Blumgart LH. Improvement in perioperative outcome after hepatic resection: analysis of 1,803 consecutive cases over the past decade. Ann Surg. 2002 Oct;236(4):397-406; discussion 406-7. doi: 10.1097/01.SLA.0000029003.66466.B3. PMID 12368667
- [Background] Poon RT, Fan ST, Lo CM, Liu CL, Lam CM, Yuen WK, Yeung C, Wong J. Improving perioperative outcome expands the role of hepatectomy in management of benign and malignant hepatobiliary diseases: analysis of 1222 consecutive patients from a prospective database. Ann Surg. 2004 Oct;240(4):698-708; discussion 708-10. doi: 10.1097/01.sla.0000141195.66155.0c. PMID 15383797
- [Background] Andreou A, Aloia TA, Brouquet A, Dickson PV, Zimmitti G, Maru DM, Kopetz S, Loyer EM, Curley SA, Abdalla EK, Vauthey JN. Margin status remains an important determinant of survival after surgical resection of colorectal liver metastases in the era of modern chemotherapy. Ann Surg. 2013 Jun;257(6):1079-88. doi: 10.1097/SLA.0b013e318283a4d1. PMID 23426338
- [Background] Sima CS, Jarnagin WR, Fong Y, Elkin E, Fischer M, Wuest D, D'Angelica M, DeMatteo RP, Blumgart LH, Gonen M. Predicting the risk of perioperative transfusion for patients undergoing elective hepatectomy. Ann Surg. 2009 Dec;250(6):914-21. doi: 10.1097/sla.0b013e3181b7fad3. PMID 19953711
- [Background] Spolverato G, Ejaz A, Kim Y, Hall BL, Bilimoria K, Cohen M, Ko C, Pitt H, Pawlik TM. Patterns of care among patients undergoing hepatic resection: a query of the National Surgical Quality Improvement Program-targeted hepatectomy database. J Surg Res. 2015 Jun 15;196(2):221-8. doi: 10.1016/j.jss.2015.02.016. Epub 2015 Mar 19. PMID 25881789
- [Background] Massicotte L, Perrault MA, Denault AY, Klinck JR, Beaulieu D, Roy JD, Thibeault L, Roy A, McCormack M, Karakiewicz P. Effects of phlebotomy and phenylephrine infusion on portal venous pressure and systemic hemodynamics during liver transplantation. Transplantation. 2010 Apr 27;89(8):920-7. doi: 10.1097/TP.0b013e3181d7c40c. PMID 20216483
- [Derived] Martel G, Baker L, Wherrett C, Fergusson DA, Saidenberg E, Workneh A, Saeed S, Gadbois K, Jee R, McVicar J, Rao P, Thompson C, Wong P, Abou Khalil J, Bertens KA, Balaa FK. Phlebotomy resulting in controlled hypovolaemia to prevent blood loss in major hepatic resections (PRICE-1): a pilot randomized clinical trial for feasibility. Br J Surg. 2020 Jun;107(7):812-823. doi: 10.1002/bjs.11463. Epub 2020 Jan 22. PMID 31965573
- [Derived] Rekman J, Wherrett C, Bennett S, Gostimir M, Saeed S, Lemon K, Mimeault R, Balaa FK, Martel G. Safety and feasibility of phlebotomy with controlled hypovolemia to minimize blood loss in liver resections. Surgery. 2017 Mar;161(3):650-657. doi: 10.1016/j.surg.2016.08.026. Epub 2016 Oct 4. PMID 27712877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phlebotomy | Control
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phlebotomy | Control | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (14) | 62 (11) | 60 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 15 | 18 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Total Intraoperative Blood Loss, by Measurement of Change in Hemoglobin Levels
Description: Intraoperative blood loss is notoriously difficult to measure. It is suggested that calculation of blood loss using preoperative and postoperative hemoglobin levels in most consistently accurate. In order to minimize the risk of bias associated with any one method of intraoperative measurement of blood loss, three methods will be used independently. In the operating room, all blood and fluid aspirated from the abdomen will be measured accurately using graduated suction containers. As well, the amount of irrigation fluid will be carefully monitored and recorded. Finally, the weight of all surgical sponges will be measured. This information will be used by the surgeon and anesthesiologist to independently visually estimate blood loss, as is commonly done in clinical practice. In parallel, intraoperative blood loss will also be calculated based on an equation.
Time Frame: 1 week prior to surgery (hemoglobin level), and day two of post-op (hemoglobin again).
Population: incomplete data
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Phlebotomy | Control
Number analyzed (Participants) | 31 | 31
mL
  Anaesthetist Estimate: number analyzed (Participants) | 30 | 31
  Anaesthetist Estimate | 862 [451 to 1187] | 872 [525 to 1314]
  Surgeon Estimate | 761 [451 to 1100] | 872 [557 to 1248]
  Calculated EBL: number analyzed (Participants) | 29 | 31
  Calculated EBL | 1116 [958 to 1526] | 1249 [778 to 1601]

2. Primary Outcome: Trial Feasibility
Description: Trial accrual
Time Frame: through study completion, an average of 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Participant Accrual: Enrolment of participants in either group (Phlebotomy or Control)
Arm/Group | Participant Accrual
Number analyzed (Participants) | 62
Participants | 62

3. Secondary Outcome: Blood Product Transfusion Rates
Time Frame: Will be measured in the operating room and in the first postoperative week
Measure: Count of Participants; unit: Participants
Arm/Group | Phlebotomy | Control
Number analyzed (Participants) | 31 | 31
Participants
  Intraoperative | 1 | 1
  Postoperative | 5 | 3
  Total | 5 | 4

4. Secondary Outcome: Perioperative Morbidity (Dindo-Clavien Grade 3b of Higher) and Mortality
Time Frame: Postoperative setting up to 30 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phlebotomy | Control
Number analyzed (Participants) | 31 | 31
Participants
  postoperative complications | 10 | 15
  Major complication | 2 | 3

5. Secondary Outcome: Changes in Physiologic Parameters (CVP)
Time Frame: Will be measured in the operating room
Population: the number analyzed in one or more rows differs from overall number analyzed due to incomplete data
Measure: Median (Inter-Quartile Range); unit: cmH2O
Arm/Group | Phlebotomy | Control
Number analyzed (Participants) | 31 | 31
cmH2O
  before transection: number analyzed (Participants) | 28 | 25
  before transection | 8 [4.5 to 9.5] | 7 [6 to 9]
  transection: number analyzed (Participants) | 25 | 22
  transection | 8 [5 to 10] | 7.5 [5 to 10]

6. Secondary Outcome: Change in Physiologic Parameters (Cardiac Index)
Time Frame: Will be measured in the operating room
Population: the number analyzed in one or more rows differs from overall number analyzed due to incomplete data
Measure: Median (Inter-Quartile Range); unit: I per min per m2
Arm/Group | Phlebotomy | Control
Number analyzed (Participants) | 31 | 31
I per min per m2
  Before transection: number analyzed (Participants) | 26 | 25
  Before transection | 3.5 [3.0 to 4.1] | 4.2 [3.2 to 5.1]
  transection: number analyzed (Participants) | 24 | 21
  transection | 3.5 [3.1 to 4.4] | 3.9 [3.1 to 5.1]

ADVERSE EVENTS:
Time Frame: adverse event data were collected for each participant for up to 30 days post surgery (intervention)
Arm/Group | Phlebotomy | Control
All-Cause Mortality (participants affected / at risk) | 2/31 | 1/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/31
Other Adverse Events (participants affected / at risk) | 8/31 | 12/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phlebotomy (N=31) | Control (N=31)
Dialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phlebotomy (N=31) | Control (N=31)
Postoperative compliations (Dindo-clavien grade I-II) (General disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT02548910/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02548910/Prot_SAP_001.pdf